CLINICAL TRIAL: NCT04548167
Title: Prolonged Cardiopulmonary Bypass Time as Predictive Factor for in Hospital Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00210; ch20Berdajs2
Record Dates: First submitted 2020-09-02; First posted 2020-09-14 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Bloodstream Infection (BSI)
Keywords: cardiovascular surgery; cardiopulmonary bypass (CPB); nosocomial infection; early bloodstream infection; postoperative septicaemia
MeSH Terms: conditions — Sepsis; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to analyse the demographics and microbiological factors concerning patients undergoing cardio surgical intervention using CPB complicated with bloodstream infection (BSI) postoperatively.

DETAILED DESCRIPTION:
Infectious complications after cardiovascular surgery, especially in operations that use cardiopulmonary bypass (CPB), is associated with significant morbidity and increase in peri-operative mortality. Prolonged CPB usage could be predictive for early bloodstream infection following cardia surgery. This study is to analyse the demographics and microbiological factors concerning patients undergoing cardio surgical intervention using CPB complicated with bloodstream infection (BSI) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing cardiac surgery

Exclusion Criteria:

* patients having active or previous endocarditis
* patients whose causative microorganism of postoperative BSI was identical to that isolated from preoperative or intraoperative samples
* patients with common skin colonized microorganisms, such as coagulase-negative Staphylococci, Viridans group Streptococci, Corynebacterium species, Bacillus species, Propionibacterium species, and Aerococcus species or Micrococcus species, which were isolated from only a single blood sample and without evidence of clinical sepsis, because contamination was considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having suffered from sepsis after cardiac surgery in a period between 2009 and 2019 will be evaluated.
Sampling Method: Probability Sample
Enrollment: 7064 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of bloodstream infection (BSI) in postoperative period (clinical evidence of sepsis with laboratory-confirmed bacteraemia from blood sample) | within 7 days after a cardiovascular surgery
  Incidence of bloodstream infection (BSI) in postoperative period (clinical evidence of sepsis with laboratory-confirmed bacteraemia from blood sample)
Extracorporeal circulation time during surgery (minutes) | one time assessment at baseline
  Extracorporeal circulation time during surgery (minutes)
In-hospital mortality (number) for patients with BSI vs those without BSI after a cardiovascular surgery | during hospital stay (usually up to 4 weeks)
  In-hospital mortality is defined as death before discharge
Surgical intervention rate (Incidence of cardiovascular re-operation) during the initial hospital stay (number) | during hospital stay (usually up to 4 weeks)
  Surgical intervention rate (Incidence of cardiovascular re-operation) during the initial hospital stay

SECONDARY OUTCOMES:
Incidence of cardiovascular events (stroke, myocardial infarction) during hospitalization | during hospital stay (usually up to 4 weeks)
  Incidence of cardiovascular events during hospitalization
Incidence of cardiovascular events (stroke, myocardial infarction) during follow-up | after hospital discharge until follow- up assessment (up to 10 years)
  Incidence of cardiovascular events (stroke, myocardial infarction) during follow-up
Incidence of cardiovascular re-operation during the follow up | after hospital discharge until follow- up assessment (up to 10 years)
  Incidence of cardiovascular re-operation during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Denis Berdajs, Prof. Dr. med., Principal Investigator — Klinik für Herzchirurgie, University Hospital Basel
Locations (1):
- Klinik für Herzchirurgie, University Hospital Basel, Basel, Switzerland